CLINICAL TRIAL: NCT02875379
Title: Clinical Comparison of Different Humidification Strategies During Noninvasive Ventilation With Helmet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Massimo Antonelli, M.D. Full Professor of Anesthesiology and Intensive Care. Head of the department of Anesthesiology and Intensive Care medicine, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 11491/15
Record Dates: First submitted 2015-07-27; First posted 2016-08-23 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Respiratory Failure
Keywords: Noninvasive Ventilation; Mechanical Ventilation
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HME (Experimental): Passive humidification with heat and moisture exchanger, Y-piece circuit.
  Interventions: Procedure: Measurements
- HH33 (Experimental): Heated humification (MR 730, Fisher & Paykel, Auckland, New Zealand), humidification chamber temperature 33°C.
  Interventions: Procedure: Measurements
- HH37 (Experimental): Heated humification (MR 730, Fisher & Paykel, Auckland, New Zealand), humidification chamber temperature 33°C.
  Interventions: Procedure: Measurements
- NoH (Experimental): Passive humidification, double tube circuit
  Interventions: Procedure: Measurements

INTERVENTIONS:
Procedure: Measurements — Measurements of respiratory mechanics and parameters, arterial blood gases and comfort

SUMMARY:
Background. Non invasive positive pressure ventilation (NIV) is among first line treatments of acute respiratory failure. Several interfaces are available for non-invasive ventilation.Despite full face and oronasal masks are more frequently used, some evidence suggests that helmets may optimize patients' comfort and NIV tolerability.

During NIV, humidification strategies (heat and moisture exchangers HME or heated humidifiers HH) may significantly affect patient's comfort and work of breathing.

Despite physiological data suggested heated humidification as the best strategy during NIV with full face masks, no differences were found in a randomized controlled study assessing the effects of HME or HH on a pragmatic clinical outcome.

However, the higher dead space (i.e. 18 L/min) and rebreathing rate observed during helmet NIV make such results not applicable to this particular setting.

The investigators designed a randomized-crossover trial to assess the effect of four humidification strategies during helmet NIV on patients with acute respiratory failure, in terms of comfort, work of breathing and patient-ventilator interaction.

Methods. All awake, collaborative, hypoxemic patients requiring mechanical ventilation will be considered for the enrollment. Hypercapnic patients (i.e.PaCO2>45 mmHg) will be excluded.

Each enrolled patient will undergo helmet NIV with all the following humidification strategies in a random order. Each period will last 60 minutes.

* Passive humidification, double tube circuit.
* Heated humification (MR 730, Fisher & Paykel, Auckland, New Zealand), humidification chamber temperature 33°C.
* Heated humification (MR 730, Fisher & Paykel, Auckland, New Zealand), humidification chamber temperature 37°C.
* Passive humidification with HME, Y-piece circuit.

Ventilatory settings (Draeger Evita xl or Evita infinity ventilators):

Pressure support ventilation; pressure support=20 cmH20; FiO2 titrated to obtain SpO2 between 92 and 98%; positive end-expiratory pressure=10 cmH2O; maximum inspiratory time 0.9 seconds; inspiratory flow trigger = 2 l/min; expiratory trigger: 30% of the maximum inspiratory flow; pressurization time=0,00 s.

Such settings will be kept unchanged during the whole study period. An oesophageal catheter will be placed and secured to measure oesophageal pressure (Pes) and gastric pressure (Pga) (Nutrivent, Italy): the reliability of the measured pressure will be confirmed with an airway occlusion test during NIV with oronasal mask. Work of breathing will be estimated with the pressure-time product (PTP) of the pleural pressure.

A pneumotachograph (KleisTek) will record flow, airway pressure, Pes and Pga on a dedicated laptop.

At the end of each cycle, the patient will be asked to rate his/her discomfort on a visual analog scale (VAS) modified for ICU patients. The level of dyspnea will be assessed with the Borg dyspnea scale.

The following parameters will be record at the end of each cycle:

Arterial pressure, heart rate, respiratory rate, SpO2, pH, PCO2, PaO2, SaO2. Airway and esophageal pressure signals will be reviewed offline to detect patient-ventilator asynchronies (ineffective efforts, double cycling, premature cycling, delayed cycling) and asynchrony index (number of asynchrony events divided by the total respiratory rate computed as the sum of the number of ventilator cycles (triggered or not) and of wasted efforts) will be computed. The trigger delay will be also measured. The pressurization and depressurization velocity will be assessed with the PTP airway index 300 and 500 (inspiratory and expiratory), as suggested by Ferrone and coworkers. The work of breathing (WOB) for each breath will be estimated by PTPes.

An hygrometer (Dimar SRL, Italy) will measure and record on a dedicated laptop Helmet temperature, relative and absolute humidity.

Primary endpoints: patient's comfort, work of breathing and asynchrony index.

Sample Sizing:

Given the physiological design of the study, the investigators did not make an a priori sample size and plan to enroll 24 patients.

DETAILED DESCRIPTION:
Background Non invasive positive pressure ventilation (NIV) is among first line treatments of acute respiratory failure. In patients with new-onset respiratory failure, NIV was showed to reduce the rate of complications and the length of ICU stay, as compared to invasive mechanical ventilation[1] Several interfaces are available for non-invasive ventilation: full face masks, oronasal masks, nasal prongs and helmets[2].

Despite full face and oronasal masks are more frequently used, some evidence suggests that helmets may optimize patients' comfort and NIV tolerability. The helmet allows patients' interaction, speech, feeding and does not limit cough. In addition, skin necrosis, gastric distension, or eye irritation are seldom observed during helmet NIV, while may be consequences of long-term treatments with face masks. [3] On the contrary, helmet NIV hampers tidal volume monitoring, is contraindicated in hypercapnic patients and requires specific ventilator settings[4]. Lastly, when compared to face masks, helmets may increase the work of breathing and worsen patient-ventilator interaction[5][6][7].

During NIV, humidification strategies (heat and moisture exchangers HME or heated humidifiers HH) may significantly affect patient's comfort and work of breathing [8][9].

Despite physiological data suggested heated humidification as the best strategy during NIV with full face masks[8][9], no differences were found in a randomized controlled study assessing the effects of HME or HH on a pragmatic clinical outcome[10].

However, the higher dead space (i.e. 18 L/min) and rebreathing rate observed during helmet NIV make such results not applicable to this particular setting.

One only study assessed the effects of a HH during helmet low-flow continuous positive airway pressure on comfort in healthy volunteers[11]. Indeed, patients suffering from acute respiratory failure may behave differently, especially in terms of minute ventilation and maximum inspiratory flow.

A recent bench study identified a better patient-ventilator interaction when helmet NIV was provided through a double tube circuit, as compared to the Y-piece system [12]. The investigators designed a randomized-crossover trial to assess the effect of four humidification strategies during helmet NIV on patients with acute respiratory failure, in terms of comfort, work of breathing and patient-ventilator interaction.

Methods Design: monocentric, randomized, cross-over trial. Each enrolled patient will undergo helmet NIV with all the following humidification strategies in a random order. Each period will last 60 minutes.

* Passive humidification, double tube circuit.
* Heated humification (MR 730, Fisher & Paykel, Auckland, New Zealand), humidification chamber temperature 33°C.
* Heated humification (MR 730, Fisher & Paykel, Auckland, New Zealand), humidification chamber temperature 37°C.
* Passive humidification with HME, Y-piece circuit.

Ventilatory settings (Draeger Evita xl or Evita infinity ventilators):

Pressure support ventilation; pressure support=20 cmH20[4]; FiO2 titrated to obtain SpO2 between 92 and 98%; positive end-expiratory pressure=10 cmH2O[4]; maximum inspiratory time 0.9 seconds; inspiratory flow trigger = 2 l/min; expiratory trigger: 30% of the maximum inspiratory flow; pressurization time=0,00 s.

Such settings will be kept unchanged during the whole study period. An oesophageal catheter will be placed and secured to measure oesophageal pressure (Pes) and gastric pressure (Pga) (Nutrivent, Italy): the reliability of the measured pressure will be confirmed with an airway occlusion test during NIV with oronasal mask[13]. Work of breathing will be estimated with the pressure-time product (PTP) of the pleural pressure[13].

A pneumotachograph (KleisTek) will record flow, airway pressure, Pes and Pga on a dedicated laptop.

At the end of each cycle, the patient will be asked to rate his/her discomfort on a visual analog scale (VAS) modified for ICU patients. The level of dyspnea will be assessed with the Borg dyspnea scale[14].

The following parameters will be record at the end of each cycle:

Arterial pressure, heart rate, respiratory rate, SpO2, pH, PCO2, PaO2, SaO2. Airway and esophageal pressure signals will be reviewed offline to detect patient-ventilator asynchronies (ineffective efforts, double cycling, premature cycling, delayed cycling) and asynchrony index (number of asynchrony events divided by the total respiratory rate computed as the sum of the number of ventilator cycles (triggered or not) and of wasted efforts) will be computed[15]. The trigger delay will be also measured. The pressurization and depressurization velocity will be assessed with the PTP airway index 300 and 500 (inspiratory and expiratory), as suggested by Ferrone and coworkers[12]. The work of breathing (WOB) for each breath will be estimated by PTPes.

An hygrometer (Dimar SRL, Italy) will measure and record on a dedicated laptop Helmet temperature, relative and absolute humidity.

End point:

Primary endpoints: patient's comfort, work of breathing and asynchrony index.

Sample Sizing:

Given the physiological design of the study, the investigators did not make an a priori sample size and planned to enroll 24 patients.

Statistical analysis Qualitative data will be expressed as number of events (%) and continuous data as mean ± standard deviation or median [Interquartile range]. Comparisons concerning qualitative variables will be performed with the Mc-Namar test. Ordinal qualitative variables or non normal quantitative variables will be compared with the Friedman's Test, the wilcoxon sum of ranks test or the Mann-Whitney test, as appropriate. All analysis will be performed applying a bilateral hypothesis. P ≤ 0.05 will be considered significant. Statistical analysis will be performed with SPSS 20.0.

ELIGIBILITY:
Inclusion Criteria:

* Awake and collaborative patients
* Age>18 years
* Need for noninvasive mechanical ventilation
* Informed consent

Exclusion Criteria:

* Cardiopulmonary resuscitation
* Haemodynamic instability
* Coma
* Asma
* Hypercapnia (paCO2>45 mmHg)
* Recent gastric or abdominal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
Comfort assessed by visual analogic scale modified for ICU patients | At the end of each 1-hour ventilation period
  Patient's comfort, assessed by visual analogic scale modified for ICU patients
Patient-ventilator asynchrony. Asynchrony index | At the end of each 1-hour ventilation period
  Asynchrony index number of asynchrony events divided by the total respiratory rate computed as the sum of the number of ventilator cycles (triggered or not) and of wasted efforts. Inspiratory trigger delay (time between the onset of patient's effort and ventilatory support). Pressurization and depressurization efficacy.
Work of breathing. Oesophageal pressure time product | At the end of each 1-hour ventilation period
  Pressure time product of the esophageal pressure (PTPes) and pressure time product of the transdiaphragmatic pressure (PTPdi)

SECONDARY OUTCOMES:
PaO2 | At the end of each 1-hour ventilation period
respiratory rate | At the end of each 1-hour ventilation period
Dyspnea | At the end of each 1-hour ventilation period
  Borg dyspnea score
Helmet humidity | At the end of each 1-hour ventilation period
Helmet temperature | At the end of each 1-hour ventilation period
PaCO2 | At the end of each 1-hour ventilation period

CONTACTS AND LOCATIONS:
Locations (1):
- General ICU, A. Gemelli hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bongiovanni F, Grieco DL, Anzellotti GM, Menga LS, Michi T, Cesarano M, Raggi V, De Bartolomeo C, Mura B, Mercurio G, D'Arrigo S, Bello G, Maviglia R, Pennisi MA, Antonelli M. Gas conditioning during helmet noninvasive ventilation: effect on comfort, gas exchange, inspiratory effort, transpulmonary pressure and patient-ventilator interaction. Ann Intensive Care. 2021 Dec 24;11(1):184. doi: 10.1186/s13613-021-00972-9. PMID 34952962